CLINICAL TRIAL: NCT04268654
Title: Trial on Ischemic Conditioning of the Gastric Conduit in Esophageal Cancer. Effects on Oxygenation and Anastomotic Leakage.
Brief Title: Ischemic Conditioning of the Gastric Conduit in Esophageal Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TIGOAL
Record Dates: First submitted 2020-02-06; First posted 2020-02-13 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-11

CONDITIONS: Esophageal Anastomotic Leak; Tissue Pressure of Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ischemic Conditioning (Experimental): Preoperative artery embolization prior to esophagectomy
  Tissue pressure of oxygen measurement in both arms by Licox system. The probe is inserted directly through the skin as a cervical drainage and it is fixed by Witzel technique in the gastric conduit. It is removed after the three measurements (intraoperatively, 24h and 48h after surgery) of the PtiO2 as a normal drainage.
  Interventions: Procedure: Preoperative Arterial Embolization
- Control (No Intervention): Surgery without previous ischemic conditioning of the gastric conduit
  Tissue pressure of oxygen measurement in both arms by Licox system. The probe is inserted directly through the skin as a cervical drainage and it is fixed by Witzel technique in the gastric conduit. It is removed after the three measurements (intraoperatively, 24h and 48h after surgery) of the PtiO2 as a normal drainage.

INTERVENTIONS:
Procedure: Preoperative Arterial Embolization — PAE will be performed by arteriographic procedure before esophageal resection surgery minimum 14 days before surgery.
  An angiogram of the celiac trunk is performed through a femoral access before and after the embolization. Embolization by coils of the left gastric artery, splenic artery and the right gastric artery is realized.
  Arms: Ischemic Conditioning

SUMMARY:
This study is a randomized clinical trial to clarify if preoperative embolization of gastric arteries can reduce the incidence of oesophagogastric leakage after an esophagectomy for esophageal cancer comparing an experimental group vs control group.

DETAILED DESCRIPTION:
In patients with infracarinal esophageal carcinoma, the surgery is a complex procedure and with a high morbidity. It consists of a subtotal esophagectomy with tubular gastroplasty and cervical esophagogastric anastomosis. The most important complication is the anastomotic leakage with a high mortality. Among the possible causes of anastomotic leakage an important factor is the impaired microcirculation in the anastomotic region after the partial devascularization of the stomach during the surgery. There are several experimental studies about the different techniques to improve this vascularization and their effects on mucosal oxygenation. There are several methods currently used for assessing tissue oxygenation. The polarographic partial pressure of oxygen (pO2) electrode has been considered as the 'gold standard' for measuring oxygen tension. This is the reason why tissue pressure of oxygen (PtiO2) will be measured by Licox® (Integra Neuroscience) system in two groups. There aren't prospective randomized controlled trials to answer these questions. For this reason the investigators propose to perform a prospective randomized controlled trial in patients underwent on this surgery, comparing two groups: one of them will be carried out a preoperative arterial embolization (PAE), and the other one will be operated directly, to demonstrate if the ischemic conditioning by PAE can reduce the incidence of anastomotic esophagogastric leakage and improve the gastric conduit oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring a esophagectomy with cervical esophagogastrostomy for esophageal cancer
* 18 or above years old
* Karnofsky>50%
* Acceptance and signing the full informed consent

Exclusion Criteria:

* Fistula tracheobronchial
* Metastatic disease
* Anatomic vascular alteration that contraindicate the embolization (congenital celiac trunk stenosis, presence of arcuate ligament, atherosclerotic stenosis, etc,..)
* Severe cardiorespiratory failure
* Refuse to collaborate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Anastomotic leakage | 90 days
  Clinic, endoscopy or computed tomography with oral contrast of dehiscence of oesophagogastric anastomosis.

SECONDARY OUTCOMES:
Tissue pressure oxygen (Ptio2) | 48 hours
  Licox oxygen monitoring system placed during the surgery in the gastric conduit. Measurements: intraoperatively and 24 hours and 48 hours after surgery.
Relation between PtiO2 and anastomotic leakage | 90 days
  We will analyse the correlation between the measurement of tissue pressure oxygen and the prevention of anastomotic leakage.
Gastric Conduit ischemia | 90 days
  Plasty ischemia when one or more of the following criteria is present:
  * Endoscopic evidence of gastric mucosa ischemia
  * Evidence in a thoracoabdominal CT with endovenous contrast
Morbidity | 90 days
  Investigator will analyse the morbidity between the two groups with the common postoperative complications: - Anastomotic leakage
  * Wound infection
  * Pulmonary complications
  * Complications related to PAE
  * Cardiologic complications
Mortality | 90 days
  Postoperative mortality has been defined as any death, regardless of cause, occurring within 30 days after surgery in or out of the hospital.
Hospital Stay | 90 days
  investigators will consider since the day of the surgery until the day the patient will be discharged from the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, VAL, Spain